CLINICAL TRIAL: NCT02398071
Title: The Effects of Breathing With a Positive Expiratory Pressure Device on The Rate of Post-exercise Recovery in Patients With COPD
Brief Title: The Effects of Positive Expiratory Pressure Breathing on The Rate of Post-exercise Recovery in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khajonsak Pongpanit (Other)
Responsible Party: Sponsor-Investigator, Khajonsak Pongpanit, Graduate School, Khon Kaen university, Khon Kaen University
Organization: Khon Kaen University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Khon Kaen University
Record Dates: First submitted 2015-03-02; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Positive Expiratory Pressure; Exercise Recovery; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEP interventon (Experimental): Participants performed 6 PEP breaths using a water pressure threshold device (BreatheMAX) with expiratory load set at 5 cmH2O
  Interventions: Device: A water pressure threshold device (BreatheMAX)
- Sham intervention (Sham Comparator): Participants performed 6 PEP breaths using a water pressure threshold device (BreatheMAX) with expiratory load set at 0 cmH2O
  Interventions: Device: A water pressure threshold device (BreatheMAX)

INTERVENTIONS:
Device: A water pressure threshold device (BreatheMAX) — BreatheMAX®, the water pressure threshold breathing device contributed in our laboratory will be used. This device is small, simple, easy to use and also inexpensive since the device is developed and manufactured in Thailand. The depth of water in the body of the device provides the flow resistance during exhalation through the inlet tube in a water cylinder.

SUMMARY:
Most daily activities involve alternating periods of exercise and rest. If recovery is slow following exercise it means that the next period of activity may be more difficult and the COPD patients becomes restricted in their daily life. Therefore, the investigators are interested to study the effectiveness and physiological effects of breathing with a PEP device during post-exercise period and hypothesize that

1. Post-exercise breathing with PEP device will increase the rate of recovery more than breathing without PEP device.
2. Post-exercise breathing with PEP device will not create harmful effects on cardiopulmonary function in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) was the 4th leading cause of morbidity and mortality worldwide in 2012 and represents an important public health challenge that is both preventable and treatable. COPD is characterized by persistent airflow limitation that is usually progressive and associated with an enhanced chronic inflammatory response in the airways and the lung to noxious particles or gases.

The pathophysiological hallmark of COPD is an expiratory air flow limitation. During exercise, increasing ventilatory demands can induce premature airway closure by forced expiration leading to air trapping and further leading to lung hyperinflation. Dynamic hyperinflation (DH) during exercise contributes to increased end expiratory lung volume (EELV), reduces inspiratory capacity (IC), and increases the mechanical load on inspiratory muscles leading to dyspnea, exercise intolerance, limited physical activity, and thus to a poor quality of life in COPD patients. In addition, abnormal lung mechanical function during dynamic hyperinflation leads to increased sensation of dyspnea, which is the disparity between respiratory drive and the respiratory mechanical response. Abnormal controls of blood chemicals and of vasculature factors also aggravate the sensation of dyspnea.

The autonomic dysfunction (AD) that occurs in the patients with COPD is evident as an inability of heart rate to reach an appropriate level during exercise (chronotropic incompetence; CI). There is also a prolonged heart rate recovery (HRR) at the end of exercise which may contribute to increase dyspnea sensations and increased mortality rate in COPD.

Expiratory flow retardation when breathing with a positive expiratory pressure (PEP) device is the one of various techniques to manage dyspnea in COPD. Most studies using a PEP device have focused on investigating the effects of PEP to reduce lung hyperinflation, reduce dyspnea, and increase exercise capacity. Only one study of Martin and Devenport, has examined the effects of PEP breathing during the recovery periods after exercise and found that following 6 minutes sub-maximal treadmill walking, 6 breath exhalation against a 10 cmH2O threshold PEP reduced dyspnea and increased HRR. Oxygen pulse saturation (SpO2) was also increased within 2 minutes although there was no statistical significant between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe COPD (both stages: FEV1/FVC < 70%, moderate stage: 50% ≤ FEV1 < 80% predicted, severe stage: 30% ≤ FEV1 < 50% predicted according to Global Initiative Obstructive Lung Disease (GOLD) guideline
* Free of exacerbations for more than 4 weeks (as defined by a change to pharmacological therapy, admission to hospital or ER or unscheduled clinic visit)
* Age between 40-70 years old
* Good communication

Exclusion Criteria:

* Musculoskeletal problems that limit mobility
* Cardiovascular disease
* Neurological or psychiatric illness
* Any other comorbidities which would affect ability to undertake exercise test

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Dyspnea rating (Rating of Perceived Breathlessness) | 5 minutes of exercise, 10 minutes of recovery periods
  collect data every minute

SECONDARY OUTCOMES:
Oxygen pulse saturation (SpO2) | 5 minutes of exercise, 10 minutes of recovery periods
  collect data every minute
End tidal carbon dioxide pressure (PETCO2) | 5 minutes of exercise and 10 minutes of recovery periods
  collect data every minute
Respiratory rate (RR) | 5 minutes of exercise, 10 minutes of recovery periods
  collect data every minute
Expiratory flow rate | 10 minutes of recovery periods
Mouth pressure | 10 minutes of recovery periods
Inspiratory capacity (IC) | at 0th, 5th minutes of exercise
Inspiratory capacity (IC) | ~1st, 10th minutes of recovery periods
Heart rate (HR) | 5 minutes of exercise, 10 minutes of recovery periods
  collect data every minute

CONTACTS AND LOCATIONS:
Overall Officials: Chulee Jones, PhD, Study Director — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Thailand; Watchara Boonsawat, PhD, Study Chair — Department of medicine, Faculty of medicine, Khon Kaen university, Thailand; David A. Jones, PhD, Study Chair — School of Healthcare Science, Faculty of Science and Engineering, Manchester Metropolitan University, United Kingdom; Khajonsak Pongpanit, MSc student, Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Thailand
Locations (1):
- School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Muang Khon Kaen, Thailand